CLINICAL TRIAL: NCT03496337
Title: Is AMPS a Responsive Tool for Assessing Change in ADL-abilities in Patients Undergoing Rehabilitation After Finger or Hand Surgery?
Brief Title: Is AMPS a Responsive Tool for Assessing Change in ADL-abilities After Finger or Hand Surgery
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 634805
Record Dates: First submitted 2018-02-06; First posted 2018-04-12 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-02

CONDITIONS: Radius Fractures; Hand Fracture; Hand Injuries
Keywords: activities of daily living; assessment of motor and process skills; validation study; responsiveness study
MeSH Terms: conditions — Radius Fractures; Hand Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of motor and process skills test — At baseline and follow-up (after 8-10 weeks) all patients are assessed with AMPS in addition to the standard test of Canadian Occupational Performance Measure (COPM) hand grip strength and joint range of motion.

SUMMARY:
The aim of the study is to assess the responsiveness of the Assessment of Motor and Process Skills (AMPS) in a population of patients undergoing rehabilitation following hand surgery, as this has not previously been investigated.

Methods: Patients are included from the department of physical and occupational therapy at Silkeborg Regional Hospital in the period November 2017 to May 2018. A total of 50 patients, who have been referred for specialized occupational therapy rehabilitation following finger or hand surgery, will be included. At baseline and follow-up (after 8 weeks) all patients are assessed with AMPS, Canadian Occupational Performance Measure (COPM), hand grip strength and joint range of motion using standardized methods. Responsiveness to change is evaluated using an anchor-based method, comparing AMPS scores with the scores on the Global Rating Scale. The area under the ROC curve will be calculated, and an area under the curve of 0.7 is considered acceptable. Convergent and discriminative validity of the AMPS will be assessed across the different instruments used. Thus the investigators expect a higher correlation between AMPS and COPM and lower correlation between AMPS and hand grip strength and range of motion.

DETAILED DESCRIPTION:
Rehabilitation following finger or hand surgery is often evaluated using only instruments assessing bodily function, e.g. hand grip strength and joint range of motion. However, considering the ICF rehabilitation framework, outcome measures should focus more on activity and participation. Furthermore, many patients requiring finger or hand surgery are still at the labor market, which underlines the importance of a valid assessment of their abilities in terms of activity and participation. This study will provide valuable knowledge in terms of whether AMPS is a valid tool for measuring improvement on these parameters in a population for which AMPS has not traditionally been used.

The aim of the study is to assess the responsiveness of the Assessment of Motor and Process Skills (AMPS) in a population of patients undergoing rehabilitation following hand surgery, as this has not previously been investigated.

Methods: Patients are included from the department of physical and occupational therapy at Silkeborg Regional Hospital in the period November 2017 to July 2018. A total of 50 patients, who have been referred for specialized occupational therapy rehabilitation following finger or hand injuries, will be included. Patients are excluded if they have movement restrictions following surgery (e.g. following surgery for tendon ruptures).

At baseline and follow-up (after 8 weeks) all patients are assessed with AMPS, Canadian Occupational Performance Measure (COPM), hand grip strength and joint range of motion using standardized methods. All test procedures are performed according to a standardized test protocol.

Statistical methods: Responsiveness to change is evaluated using an anchor-based method, comparing AMPS scores with the scores on the Global Rating Scale. The area under the ROC curve will be calculated, and an area under the curve of 0.7 is considered acceptable. Convergent and discriminative validity of the AMPS will be assessed across the different instruments used. Thus a higher correlation between AMPS and COPM and lower correlation between AMPS and hand grip strength and range of motion is expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for occupational therapy rehabilitation at Silkeborg Regional Hospital following surgery of the forearm, wrist, hand or fingers.

Exclusion Criteria:

* Patients who cannot perform rehabilitation due to movement restrictions following surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are included from the department of physical and occupational therapy at Silkeborg Regional Hospital in the period November 2017 to May 2018. A total of 50 patients, who have been referred for specialized occupational therapy rehabilitation following finger, hand, wrist or forearm surgery, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in "Assessment of motor and process skills (AMPS)" from baseline to 8 weeks | Measured at baseline and 8 weeks after baseline
  The Assessment of Motor and Process Skills (AMPS) is an observational assessment that allows for the simultaneous evaluation of motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living. After an initial interview with the patient, the rater selects a subset of 3-5 ADL tasks from a list of standardized tasks that are described in the AMPS manual (e.g. fetching a drink from the fridge, folding laundry, preparing a sandwich). The tasks selected must be relevant and meaningful to the patient, and consist of tasks that he/she once knew how to perform. The tasks must be challenging to the patient. From this subset of tasks, the client then selects 2-3 tasks to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Regionshospitalet Silkeborg
Locations (1):
- Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No